CLINICAL TRIAL: NCT06660927
Title: A Study on the Safety and Efficacy of the G-iliac Iliac Bifurcation Stent Graft System for Endovascular Repair of Common Iliac Artery Aneurysms
Brief Title: The Study on the Safety and Efficacy of the G-iliac Iliac Bifurcation Stent Graft System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 50CT(CN) L-01
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Common Iliac Artery Aneurysm
Keywords: Lifetech; Iliac Bifurcation Stent Graft System; Endovascular Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular Treatment of Patients with Common Iliac Artery Aneurysms (Experimental): Endovascular Treatment of Patients with Common Iliac Artery Aneurysms Using the Iliac Bifurcation Stent Graft System
  Interventions: Device: liac Bifurcation Stent Graft System

INTERVENTIONS:
Device: liac Bifurcation Stent Graft System — to evaluate the Safety and Efficacy of the G-iliac Iliac Bifurcation Stent Graft System for Endovascular Repair of Common Iliac Artery Aneurysms(CIAA)

SUMMARY:
The objective of this study is to evaluate the Safety and Efficacy of the G-iliac Iliac Bifurcation Stent Graft System for Endovascular Repair of Common Iliac Artery Aneurysms(CIAA).

DETAILED DESCRIPTION:
The physician shall strictly follow the clinical study protocol and shall not deviate from or substantially change the protocol. However, in case of emergency such as immediate risk to the subjects, which needs tobe eliminated immediately, it may be reported in written form afterwards. During the course of the study,documents such as amendments to the clinical study protocol and informed consent, requests for deviation,and resumption of the suspended clinical study shall be subject to the written approval of the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone implantation of the iliac bifurcation stent graft system;
* Patients with complete medical records

Exclusion Criteria:

* Patients with ruptured aortic aneurysm;
* Patients with infected or mycotic aortic aneurysm;
* Patients with connective tissue diseases, such as systemic lupus erythematosus, Marfan syndrome, Ehlers-Danlos syndrome, or Behcet's disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Major Adverse Events (MAE) within 30 Days postoperatively. | within 30 Days postoperatively
  Major Adverse Events (MAE) are defined as follows: all-cause mortality related to iliac artery aneurysms associated with the surgery or device, myocardial infarction, renal failure, respiratory failure, paraplegia, stroke, and intestinal ischemia.
he patency rate of internal iliac artery (IIA) at 12 months postoperatively | at 12 months postoperatively
  The patency rate of internal iliac artery (IIA) defined as blood flow without occlusion maintained through the device without intervention

SECONDARY OUTCOMES:
The incidence of conversion to open surgery or secondary interventional procedures due to iliac artery aneurysms before discharge and at 12 months postoperatively. | before discharge and at 12 months postoperatively
  Notes: Due to the patient's condition, the surgeon's choice of staged reconstruction does not constitute a secondary surgical intervention.
Device-related adverse events before discharge and at 12 months postoperatively | before discharge and at 12 months postoperatively.
  Device-related adverse events are those situations that are ultimately determined to be definitely related, possibly related, or indeterminate with respect to the study device.
The incidence of malfunction before discharge and at 12 months postoperatively. | before discharge and at 12 months postoperatively.
  Malfunction means the failure of a device to meet its performance specifications or otherwise perform as intended.Performance specifications include all claims made in the labeling for the device. The intended performance of a device refers to the intended use for which the device is labeled or marketed.
Incidence rate of Type I/III endoleak caused by the iliac bifurcation system that necessitate reintervention before discharge and at 12 months postoperatively. | before discharge and at 12 months postoperatively.
  Type I endoleak, also known as peri-graft endoleak or graft-related endoleak, refers to the leakage caused by the inability of the stent graft to tightly adhere to the autologous vessel, leading to continuous blood flow into the aneurysm sac. This includes proximal and distal Type I endoleaks. Type III endoleak refers to the leakage caused by the inability of the stent graft's own connectors to tightly adhere or the rupture of the artificial vessel, which results in continuous blood flow into the aneurysm sac.
The immediate technical success during intraoperative procedures. | during intraoperative procedures
  immediate technical success refers to successful delivery of the stent to the intended location by the delivery system, successful deployment of the stent, and safe removal of the delivery system. Additionally, angiography should show unobstructed blood flow within the stent, with no stent kinking, folding, narrowing, or occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: hongpeng zhang, Professor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China